CLINICAL TRIAL: NCT03112486
Title: Predicting Neurological Outcome Following Out of Hospital Cardiac Arrest (OHCA) by Quantitative Measurement of Serial Serum Biomarkers of Brain Injury.
Brief Title: Out-of-hospital Cardiac Arrest (OHCA) Biomarkers
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201700133
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Neurological Outcome; Cardiac Arrest; Out-Of-Hospital Cardiac Arrest; Brain Anoxia Ischemia; Hypoxia, Brain; Hypoxia-Ischemia, Brain; Cardiac Arrest With Successful Resuscitation; Cardiac Arrest, Out-Of-Hospital; Brain Injuries
Keywords: out-of-hospital cardiac arrest; neurological outcome; prognostication; cerebral performance category; hypoxic-ischemic brain injury; biomarkers
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Hypoxia-Ischemia, Brain; Hypoxia, Brain; Brain Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiac Arrest cohort: adult patients (≥ 18 years of age) with non-traumatic out of hospital cardiac arrest
  Interventions: Procedure: blood draw
- Control cohort: matched control population will include hemodynamically stable patients who present to the ED with chest pain that is not of cardiac etiology (non-traumatic chief complaints).
  Interventions: Procedure: blood draw

INTERVENTIONS:
Procedure: blood draw — Blood draws will be collected via venipuncture or IV at hours 0, 6, 12, 18, 24, 48, 72, 96, 120, 144 (10 draws total). Each draw would be approximately 20 mL of blood (but no less than 10 mL).

SUMMARY:
Few early prognostic indicators are currently available for patients' families and clinicians following out of hospital cardiac arrest (OHCA), and blood biomarkers may be of prognostic value in these cases. Brain tissue is highly dependent upon aerobic respiration, and oxygen deprivation result in irreversible neuronal cell injury. Peptides released into the blood by injured neuronal cells can be measured to estimate degree of injury, and potentially predict long term neurological outcome.

DETAILED DESCRIPTION:
Aggressive treatment for patients with out-of-hospital cardiac arrest (OHCA) can result in return of spontaneous circulation (ROSC). However, prognosis for these patients remains poor, with low rates of survival to hospital admission and low rates of survival to hospital discharge. Furthermore, due to the exquisite sensitivity to hypoxic injury of neural tissue (dependent on aerobic respiration) relative to that of cardiac muscle, patients for whom ROSC can be obtained often suffer devastating neurological injury, with potential poor long-term neurological outcome. In some ischemic processes, for example, myocardial infarction, rapid measurement of cardiac biomarkers (e.g. Troponin isoform) is invaluable to current diagnosis and management. However, with regards to ischemic brain injury, there is currently no rapid, definitive diagnostic test to prognosticate outcome in OHCA. Biomarkers measurable in blood would have vital applications in prognosis and clinical research of neurological outcome in OHCA.

Other groups have studied the neurological predictive values of biomarkers after OHCA. A variety of proteins including S100B, neuron-specific enolase, and G-FAP, co-peptin, Tau, neurofilament light/ heavy chain, and secretoneurin have been proposed as potential biomarkers of neurological outcome at OHCA. Unfortunately, many of these have been shown to have several drawbacks. For example, some lack specificity due to being released during resuscitation (e.g., S100B is found extracerebrally in muscle, adipocytes, and chondrocytes, creating a confounding factor in CA patients receiving chest compressions). Others have lacked sufficient sensitivity in the prognosticating of neurological outcome (ref). Furthermore, there is a paucity of human studies in cardiac arrest on newer biomarkers that have been studied in other acute brain injury disease processes that could potentially serve as candidate biomarkers predicting neurological outcome at post cardiac arrest hypoxic brain injuries. Biomarkers such as UCH-L1, SBDP, and MBP have not been studied in a OHCA cohort.

The Investigator therefore propose a prospective, observational study in which the investigator will incorporate a minimally invasive and minimal risk measurement of blood biomarkers at time of ROSC. This would be done by drawing blood at ROSC (0-59mins), and additional blood draws at hours 6, 12, 18, 24, 48, 72, and on day 4, 5, and 6. The Investigator will then determine whether biomarker levels correlates with survival to hospital admission, survival to hospital discharge, and functional neurologic outcome at discharge and at 6 months. The Investigator intend to sample patients that present to the emergency department with non-CA chest pain in our study as well, which will allow us to draw stable inferences.

ELIGIBILITY:
Inclusion Criteria:

- >18 years old

Study cohort:

* Non-traumatic out of hospital cardiac arrest
* Control cohort:
* Chest pain of non-cardiac etiology

Exclusion Criteria:

Both cohorts:

* Females of child bearing age with positive pregnancy test
* Neurodegenerative disease or other neurological disorder (dementia, Parkinson's disease, multiple sclerosis, seizure disorder, or brain tumours)
* History of neurosurgery within the last 30 days Acute brain injury within the last 30 days (ischemic/ haemorrhagic stroke, traumatic brain injury) Subject is anemic OR donated blood within the last 8 weeks OR has a hematological disorder that requires transfusions Subject has history of liver failure OR renal failure

Study cohort:

Advanced directives against resuscitation Traumatic cardiac arrest In hospital cardiac arrest Failure to attain ROSC + visible signs of death (livor mortis, rigor mortis)

Control cohort:

EKG changes: New ST-elevation consistent with myocardial infarction NSTEMI Hemodynamically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include all adult patients (≥ 18 years of age) with non-traumatic out of hospital cardiac arrest. Exclusions will include patients with advanced directives precluding resuscitation, traumatic cardiac arrest, and irreversible signs of death (e.g. rigor mortis). A matched control population will include hemodynamically stable patients who present to the ED with chest pain that is not of cardiac etiology (non-traumatic chief complaints). Blood draws in this cohort will be collected as per protocol and will end upon the termination of medical care or as per protocol - whichever is of the least duration.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 1 year
  Higher blood biomarker levels will correlate with reduced rate of survival to hospital admission, survival to hospital discharge, and 6-month survival.

SECONDARY OUTCOMES:
Functional neurological outcome at discharge | 1 year
  Higher blood biomarker levels will correlate with higher degree of neurological impairment as measured by Cerebral Performance Category.
Functional neurological outcome at 6 months after discharge | 1 year
  Higher blood biomarker levels will correlate with higher degree of neurological impairment as measured by Cerebral Performance Category.

OTHER OUTCOMES:
Influence of renal and liver disease on blood biomarker(s) level post-OHCA | 1 year
  Renal and liver disease may affect levels of protein biomarkers after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Tyndall, MD, MPH, Principal Investigator — Chairman Department Emergency Medicine
Locations (1):
- Univeristy of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Sasson C, Hegg AJ, Macy M, Park A, Kellermann A, McNally B; CARES Surveillance Group. Prehospital termination of resuscitation in cases of refractory out-of-hospital cardiac arrest. JAMA. 2008 Sep 24;300(12):1432-8. doi: 10.1001/jama.300.12.1432. PMID 18812534
- [Background] Chan PS, McNally B, Tang F, Kellermann A; CARES Surveillance Group. Recent trends in survival from out-of-hospital cardiac arrest in the United States. Circulation. 2014 Nov 18;130(21):1876-82. doi: 10.1161/CIRCULATIONAHA.114.009711. PMID 25399396
- [Background] Neumar RW, Nolan JP, Adrie C, Aibiki M, Berg RA, Bottiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT Jr, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Vanden Hoek T. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A consensus statement from the International Liaison Committee on Resuscitation (American Heart Association, Australian and New Zealand Council on Resuscitation, European Resuscitation Council, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Asia, and the Resuscitation Council of Southern Africa); the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; and the Stroke Council. Circulation. 2008 Dec 2;118(23):2452-83. doi: 10.1161/CIRCULATIONAHA.108.190652. Epub 2008 Oct 23. No abstract available. PMID 18948368
- [Background] Laver S, Farrow C, Turner D, Nolan J. Mode of death after admission to an intensive care unit following cardiac arrest. Intensive Care Med. 2004 Nov;30(11):2126-8. doi: 10.1007/s00134-004-2425-z. Epub 2004 Sep 9. PMID 15365608
- [Background] Moulaert VR, Verbunt JA, van Heugten CM, Wade DT. Cognitive impairments in survivors of out-of-hospital cardiac arrest: a systematic review. Resuscitation. 2009 Mar;80(3):297-305. doi: 10.1016/j.resuscitation.2008.10.034. Epub 2008 Dec 30. PMID 19117659
- [Background] Lim C, Verfaellie M, Schnyer D, Lafleche G, Alexander MP. Recovery, long-term cognitive outcome and quality of life following out-of-hospital cardiac arrest. J Rehabil Med. 2014 Jul;46(7):691-7. doi: 10.2340/16501977-1816. PMID 24849762
- [Background] Larsson IM, Wallin E, Rubertsson S, Kristofferzon ML. Health-related quality of life improves during the first six months after cardiac arrest and hypothermia treatment. Resuscitation. 2014 Feb;85(2):215-20. doi: 10.1016/j.resuscitation.2013.09.017. Epub 2013 Oct 2. PMID 24096198
- [Background] Pusswald G, Fertl E, Faltl M, Auff E. Neurological rehabilitation of severely disabled cardiac arrest survivors. Part II. Life situation of patients and families after treatment. Resuscitation. 2000 Nov;47(3):241-8. doi: 10.1016/s0300-9572(00)00240-9. PMID 11114453
- [Background] Sandroni C, Cavallaro F, Callaway CW, Sanna T, D'Arrigo S, Kuiper M, Della Marca G, Nolan JP. Predictors of poor neurological outcome in adult comatose survivors of cardiac arrest: a systematic review and meta-analysis. Part 1: patients not treated with therapeutic hypothermia. Resuscitation. 2013 Oct;84(10):1310-23. doi: 10.1016/j.resuscitation.2013.05.013. Epub 2013 Jun 27. PMID 23811182
- [Background] Sandroni C, Cavallaro F, Callaway CW, D'Arrigo S, Sanna T, Kuiper MA, Biancone M, Della Marca G, Farcomeni A, Nolan JP. Predictors of poor neurological outcome in adult comatose survivors of cardiac arrest: a systematic review and meta-analysis. Part 2: Patients treated with therapeutic hypothermia. Resuscitation. 2013 Oct;84(10):1324-38. doi: 10.1016/j.resuscitation.2013.06.020. Epub 2013 Jul 3. PMID 23831242
- [Background] Sandroni C, Geocadin RG. Neurological prognostication after cardiac arrest. Curr Opin Crit Care. 2015 Jun;21(3):209-14. doi: 10.1097/MCC.0000000000000202. PMID 25922894
- [Background] Perkins GD, Jacobs IG, Nadkarni VM, Berg RA, Bhanji F, Biarent D, Bossaert LL, Brett SJ, Chamberlain D, de Caen AR, Deakin CD, Finn JC, Grasner JT, Hazinski MF, Iwami T, Koster RW, Lim SH, Huei-Ming Ma M, McNally BF, Morley PT, Morrison LJ, Monsieurs KG, Montgomery W, Nichol G, Okada K, Eng Hock Ong M, Travers AH, Nolan JP; Utstein Collaborators. Cardiac arrest and cardiopulmonary resuscitation outcome reports: update of the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest: a statement for healthcare professionals from a task force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia); and the American Heart Association Emergency Cardiovascular Care Committee and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Circulation. 2015 Sep 29;132(13):1286-300. doi: 10.1161/CIR.0000000000000144. Epub 2014 Nov 11. PMID 25391522